CLINICAL TRIAL: NCT04616976
Title: Efficiency of Convalescent Plasma Therapy in Management of Critically Ill Patients With COVID-19: a Matched Case-control Study
Brief Title: COVID-19 With Convalescent Plasma
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, Dr, Southeast University, China
Other Study IDs: COVID-19 convalescent plasma
Record Dates: First submitted 2020-11-01; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: COVID-19 Convalescent Plasma Treatment
Keywords: convalescent plasma therapy; COVID-19; mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- convalescent plasma therapy group: the patients received convalescent plasma therapy
  Interventions: Biological: convalescent plasma
- Control group: the patients with similar situation without convalescent plasma therapy

INTERVENTIONS:
Biological: convalescent plasma — convalescent plasma was get from the patients who recovery from COVID-19
  Groups: convalescent plasma therapy group

SUMMARY:
To clarify the effects of convalescent plasma therapy on SARS-CoV-2 negative conversion rate during hospital stay and 28-day mortality of severe and life-threatening COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age;
2. laboratory-confirmed diagnosis of COVID-19;
3. respiratory failure requiring advanced respiratory support (i.e. high flow nasal cannula[HFNC], noninvasive mechanical ventilation [NIV], and invasive mechanical ventilation [IMV]).

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with COVID-19 who were admitted to ICUs of the participating hospitals between January 1 to February 29, 2020 were screened.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  the mortality from ICU admission to 28 days after admission

SECONDARY OUTCOMES:
SARS-CoV-2 negative conversion rate | up to 60 days
  SARS-CoV-2 viral shedding

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan C, Chen H, Xie J, Huang Y, Yang Y, Du B, Qiu H. The Efficiency of Convalescent Plasma Therapy in the Management of Critically Ill Patients Infected With COVID-19: A Matched Cohort Study. Front Med (Lausanne). 2022 Jun 16;9:822821. doi: 10.3389/fmed.2022.822821. eCollection 2022. PMID 35783610